CLINICAL TRIAL: NCT01343563
Title: Trigeminal Nerve Stimulation for Depression: Dose Finding
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Ian A. Cook, M.D., Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-000480; 10-000480 (Other: UCLA Medical IRB 3)
Record Dates: First submitted 2011-04-05; First posted 2011-04-28 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Depression
Keywords: Depression; Major Depressive Disorder (MDD); EEG; Trigeminal Nerve Stimulation
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low frequency to High (Active Comparator): For the first six weeks, subjects randomized to this group will receive low frequency stimulation. At the six week point, the low frequency group subjects will be crossed over to high frequency for the remaining six weeks.
  Interventions: Procedure: Trigeminal Nerve Stimulation
- High frequency (Active Comparator): Subjects randomized to this group will receive high frequency stimulation for the entire 12 weeks of the first phase of this study.
  Interventions: Procedure: Trigeminal Nerve Stimulation

INTERVENTIONS:
Procedure: Trigeminal Nerve Stimulation — External trigeminal nerve stimulation (TNS) as an adjunctive treatment added onto antidepressant medications.

SUMMARY:
This study will aim to examine the use of external trigeminal nerve stimulation (TNS) as an adjunctive treatment for adults with major depressive disorder (MDD) when added onto antidepressant medications. Our primary objective is the examination of two different "doses" of TNS, in terms of pulse frequency.

To accomplish our specific aims, the investigators will test the following specific hypotheses:

1. Subjects will show greater improvement in ratings of mood and other symptoms of depression during the six-week of high frequency stimulation than during low frequency stimulation periods.
2. Subjects will show greater improvement after 12 weeks of high frequency stimulation than after six weeks of high frequency stimulation.
3. Subjects will show improvement in ratings of life functional capacity and quality of life with TNS.
4. Subjects will report the TNS treatments to be acceptable in terms of side effects and burden of using the device.
5. Subjects will show significant differences in regional brain function at the end of the high frequency stimulation period compared with baseline, and significant differences between high and low frequency stimulation conditions.

DETAILED DESCRIPTION:
A total of 20 subjects with Major Depressive Disorder (MDD), ages 18 to 65, will be consented and join this project at UCLA.

The project has two phases: a 12 week treatment phase and a 6 month follow-up phase. In the first phase, a double-blind one-way cross-over design will allow us to compare the clinical and physiologic responses to TNS at two frequencies of stimulation, "high" (~120 Hz) and "low " (~20 Hz). Subjects will be randomized to start a six week period at either high or low frequency stimulation (n=10 in each); both subjects and the staff who interact with them will be blinded to assignment, and a separate member of the team will program the device settings. At the six week point, the low frequency group subjects will be crossed over to high frequency, while the high frequency group will continue at high frequency. At the end of the 12 weeks, the TNS systems will be returned and the adjunctive treatment will end. All subjects will be followed for another six months with monthly telephone calls to monitor symptoms or changes in treatment that would signal a return of symptoms. The primary endpoint is the change in depression severity for the two groups at the week 6 visit.

ELIGIBILITY:
Inclusion Criteria

1. Outpatients with non-psychotic, unipolar Major Depressive Disorder assessed via the MINI structured interview
2. A score of ≥ 14 on the HAM-D17 with Item 1 (depressed mood) ≥ 2
3. A history of treatment failure with at least one adequate trial of an antidepressant over the previous 6 weeks, with no change in antidepressant medication or dose within the previous 6 weeks, and ongoing use of at least one antidepressant (which will continue during participation in the study)
4. Age range: 18 to 65 years old.
5. Patients with suicidal ideation are eligible only if the thoughts of death or of life not being worth living are not accompanied by a plan or intention for self-harm.

Exclusion Criteria

1. Patient is mentally or legally incapacitated, unable to give informed consent.
2. Patients with psychosis (psychotic depression, schizophrenia, or schizoaffective diagnoses (lifetime)); bipolar disorder (lifetime); dementia (lifetime); delirium or any substance abuse disorder within the past 6 months; eating disorder within the past year; obsessive-compulsive disorder (lifetime); post-traumatic stress disorder within the past year; acute risk for suicide or self-injurious behavior. Patients with diagnostic uncertainty or ambiguity (e.g. rule-out pseudodementia of depression) will be excluded.
3. Patients with exposure to ECT or VNS within the past 6 months.
4. Past history of skull fracture; cranial surgery entering the calvarium; space occupying intracranial lesion; stroke, CVA, or TIAs; cerebral aneurysm; Parkinson's or Huntington's disease; or Multiple Sclerosis.
5. current pregnancy, breast feeding, plans to become pregnant in the 12-week treatment phase of the study, or not using a medically accepted means of contraception.
6. Other medical contraindications to any of the study procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale 17 score | baseline, week 6, week 12

SECONDARY OUTCOMES:
Change in life functional capacity and quality of life scales | baseline, week 6, week 12
  Life functional capacity and quality of life scales include: Short-form Health Survey-36 Item and Quality of Life Enjoyment and Satisfaction Questionnaire
Changes in Regional Brain Function | baseline, week 6, week 12
  As measured by qualitative electroencephalographic (QEEG) recordings
Changes in vital signs recordings | At every visit for 12 weeks
  Autonomic function (i.e. pulse and blood pressure) are monitored for 30 mins of stimulation at baseline, week 6, and week 12. Resting vital signs are recorded for each visit.
Changes in Safety Assessment Measures | At every visit for 12 weeks
  Safety Assessment measures will be administered at each visit and include: Survey of Acceptability of TNS, Systematic Assessment for Treatment Emergent Events-Systematic Inquiry (SAFTEE-SI), and Frequency, Intensity, and Burden of Side Effects Scale (FIBSER)

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Cook, MD, Principal Investigator — Semel Institute for Neuroscience and Human Behavior
Locations (1):
- Semel Institute for Neuroscience and Human Behavior at UCLA, Los Angeles, California, United States